CLINICAL TRIAL: NCT01540292
Title: Mesenchymal Stem Cell Therapy for the Treatment of Severe or Refractory Inflammatory and/or Autoimmune Disorders
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Yves Beguin, Professor, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJT1123
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Mesenchymal Stem Cell; Cell therapy; Allogeneic; Inflammatory disorders; Autoimmune disorders
MeSH Terms: conditions — Crohn Disease; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MSC (Experimental): Patients with Crohn's disease (refractory or intolerant to conventional therapies) treated with 2 successive injections of 1.5-2.0 x 10E6 allogenic MSC/kg BW at baseline and 4 weeks later.
  Interventions: Biological: Mesenchymal Stem Cells (MSC)

INTERVENTIONS:
Biological: Mesenchymal Stem Cells (MSC) — MSC (1.5-2 cells/kg BW) IV injection, twice at 4 weeks apart

SUMMARY:
This project aims to assess safety and efficacy of allogeneic Mesenchymal stem Cell (MSC) in Crohn's disease refractory or intolerant to conventional therapies. Twenty patients with active refractory Crohn's disease defined by a Crohn's Disease Activity Index (CDAI) > 220 despite conventional treatment will be included over 4 years in this phase I-II trial. This will be a pilot open label trial. Patients will be treated with 2 successive injections of allogeneic MSC at baseline and 4 weeks later. Patients will be followed up at weeks 2, 4, 8 and 12.

DETAILED DESCRIPTION:
1. Collection and expansion of MSC Bone marrow collection and MSC expansion cultures will be carried out at the Laboratory of Cell and Gene Therapy (LTCG) at the University of Liège. Bone marrow (50 ml) will be collected from unrelated donors under local anesthesia, mononuclear cells will be isolated, and cultured for a total of about 4 weeks. After a sufficient number of passages, the cells will be harvested, washed and frozen.
2. MSC injections MSC will be thawed and diluted at the Laboratory of Cell and Gene Therapy (LTCG), transported to the hospital ward and injected intravenously within 1 hour of thawing through a central catheter (when available) or a good peripheral vein. A dose of 1.5 - 2.0 x 106/kg recipient MSC should be ideally administered at each infusion. MSC will be infused even if the number of post-thaw cells is lower than that. Patients with Crohn's disease will receive two injections of allogenic MSC 4 weeks apart (week 0 and 4).
3. Patients Follow up

3.1. Quality controls of MSC products Quality controls of MSC product will include microscopy, nucleated cell count and differential, cell viability testing, microbiology testing (including standard virology, bacterial culture and detection of mycoplasmal enzymes by bioluminescence, endotoxin testing, karyotype and FACS analysis (cells must be positive for :CD90 > 70%,CD105 > 70 %,CD73 > 70 %; and negative for :CD14 < 5%,CD34 < 5%, CD45 < 5%, CD3 < 1%).

3.2. Toxicities of cell infusions: Potential toxicities associated with MSC infusions will be carefully monitored per the institution's standards and documented on the infusion report and/or the SAE report form. No dosage modifications are scheduled. In case of severe reaction to the first MSC infusion, the second infusion will not be performed.

3.3. Clinical data The following parameters will be followed at baseline as well as at week 2, 4, 8 and 12 : CDAI level, CRP levels, fecal calprotectin levels. In addition, duration of hospitalization, infections, any other serious complication, and eath and survival will be recorded.

3.4. Immunologic data: Immune function in the patient will be monitored at baseline and appropriate intervals: nucleated cell count and differential; FACS analysis with determination of the % cells (on total WBC) with the markers :CD3+, CD4+, CD8+, CD19+, CD45RA+, CD45RO+, CD56+, CD3+CD4+, CD3+CD8+; CD3+CD56+; CD4+CD45RA+, CD4+CD45RO+; CD3-CD56+; regulatory T-cell (Treg) levels; immunoglobulin levels, Vβ repertoire of T lymphocytes; TRECs quantification in T lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old
* Crohn's disease affecting terminal ileum, colon or both with diagnosis confirmed according to Lennard Jones criteria
* Clinically active disease with a CDAI between 220 and 450 and biologically active disease with a CRP > 5 mg/l and/or fecal calprotectin > 150 microg/g
* Resistance or intolerance to mesalazine, steroids, purine analogues, methotrexate, infliximab and adalimumab
* Adequate venous access (central catheter or good peripheral veins)
* Willingness to sign the informed consent and enter the clinical trial

Exclusion Criteria:

* Any condition not fulfilling inclusion criteria
* Indication for surgery
* Symptomatic stricture
* Undrained perianal or intraabdominal abscess
* Change in mesalazine dosage within the last 4 weeks, change in steroid dosage within the last two weeks, change in immunosuppressant dosage within the last 3 months, use of anti-TNF treatment within the last two months
* HIV positive
* Uncontrolled infection, arrhythmia or hypertension
* Terminal organ failure:

  * Renal: anuria, serious fluid overload, GFR < 30 ml/min, dialysis;
  * Pulmonary: DLCO < 35% and/or receiving supplementary continuous oxygen;
  * Hepatic: Fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease;
  * Cardiac: Symptomatic coronary artery disease or other cardiac failure requiring therapy; ejection fraction < 35%; uncontrolled arrhythmia, uncontrolled hypertension

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical Response Rate | at week 8
  To assess clinical response rate defined by a 100 points decrease in Crohn's Disease Activity Index.

SECONDARY OUTCOMES:
Clinical Response | at week 2, 4, 8 and 12.
Remission | at week 2, 4, 8 and 12.
  Remission, defined by Crohn's Disease Activity Index <150
Crohn's Disease Activity Index Level | at week 2, 4, 8 and 12.
C-reactive Protein levels | at week 2, 4, 8 and 12.
  C-reactive Protein measured in blood.
Fecal calprotectin levels | at week 2, 4, 8 and 12.
  Fecal calprotectin measured in stool samples
Immune modulation investigation | at week 12.
  The following parameters will be taken in account.
  * Nucleated cell count and differential on an automated cell counter;
  * FACS analysis with determination of the % cells (on total WBC) with the markers :
    * CD3+, CD4+, CD8+, CD19+, CD45RA+, CD45RO+, CD56+
    * CD3+CD4+, CD3+CD8+; CD3+CD56+;
    * CD4+CD45RA+, CD4+CD45RO+;
    * CD3-CD56+.
  * Regulatory T-cell (Treg) levels;
  * Immunoglobulin levels (baseline and week 12);
  * Vβ repertoire of T lymphocytes (baseline and week 12);
  * TRECs quantification in T lymphocytes (baseline and week 12).
Incidence of infections | by week 12

CONTACTS AND LOCATIONS:
Overall Officials: Yves Beguin, MD, PhD, Study Chair — CHU-ULg; Edouard Louis, MD, PhD, Principal Investigator — CHU-ULg
Locations (1):
- University Hospital Liège, Liège, Belgium